CLINICAL TRIAL: NCT00359905
Title: Evaluation of the Efficacy and Safety of Silodosin vs. Tamsulosin and Placebo in the Treatment of the Signs and Symptoms of BPH. Multicentre, Randomised, Double-Blind, Controlled Trial With an Optional Long-Term, Open-Label Extension Phase.
Brief Title: Evaluation of the Efficacy and Safety of Silodosin in the Treatment of the Signs and Symptoms of BPH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RECORDATI GROUP (Industry)
Responsible Party: Senior Clinical Project Leader, Recordati Industria Chimica e Farmaceutica S.p.A.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KMD3213-IT-CL 0215
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign prostatic hyperplasia; alpha-blockers
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — silodosin; Tamsulosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Silodosin (Experimental)
  Interventions: Drug: Silodosin
- Tamsulosin (Active Comparator)
  Interventions: Drug: Tamsulosin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Silodosin — 8 mg daily for 12 weeks
  Other Names: KMD3213
  Arms: Silodosin
Drug: Tamsulosin — 0.4 mg daily for 12 weeks
  Other Names: Omnic
  Arms: Tamsulosin
Drug: Placebo — once daily for 12 weeks
  Arms: Placebo

SUMMARY:
A new drug for the treatment of benign prostatic hyperplasia is compared with placebo and tamsulosin (a drug belonging to the same therapeutic class) for to determine if it is safe and effective (the first phase of the study lasts approximately 18 weeks) and then is used for another 9 months to determine its long-term safety.

DETAILED DESCRIPTION:
This is a multi-centre, double-blind, placebo and active controlled, parallel 12 week treatment trial in men with signs and symptoms of benign prostatic hyperplasia, followed by a 9 month open-label phase. The following procedures are used: physical exams, electrocardiograms, clinical laboratory tests, vital signs, the International Prostate Symptom Score, maximum urine flow rate, adverse events, concomitant medications, quality of life and compliance. 93 centres in 11 European countries (Finland, France, Germany, Italy, Netherlands, Poland, Romania, Russia, Spain, Ukraine, UK) will be involved

ELIGIBILITY:
Inclusion Criteria:

* Males in good general health and at least 50 years of age, with symptoms of moderate to severe Benign Prostatic Hyperplasia

Exclusion Criteria:

* Medical conditions that would confound the efficacy evaluation
* Medical conditions in which it would be unsafe to use an alpha-blocker
* Use of concomitant drugs that would confound the efficacy evaluation
* Use of concomitant drugs that would be unsafe with this alpha-blocker

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1228 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Change in baseline total score on the International Prostate Symptom Score | 12 weeks

SECONDARY OUTCOMES:
Change in baseline obstructive subscore of the International Prostate Symptom Score; | 12 weeks
change in baseline irritative subscore of the International Prostate Symptom Score; | 12 weeks
change in baseline maximum urine flow rate; | 12 weeks
safety | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Re Chapple, BSc MD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust, Royal Hallamshire Hospital
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Royal Hallamshire Hospital, Sheffield, United Kingdom

REFERENCES:
- [Derived] Osman NI, Chapple CR, Tammela TL, Eisenhardt A, Oelke M. Open-label, 9-month extension study investigating the uro-selective alpha-blocker silodosin in men with LUTS associated with BPH. World J Urol. 2015 May;33(5):697-706. doi: 10.1007/s00345-015-1519-2. Epub 2015 Feb 25. PMID 25712312
- [Derived] Chapple CR, Montorsi F, Tammela TL, Wirth M, Koldewijn E, Fernandez Fernandez E; European Silodosin Study Group. Silodosin therapy for lower urinary tract symptoms in men with suspected benign prostatic hyperplasia: results of an international, randomized, double-blind, placebo- and active-controlled clinical trial performed in Europe. Eur Urol. 2011 Mar;59(3):342-52. doi: 10.1016/j.eururo.2010.10.046. Epub 2010 Nov 10. PMID 21109344